CLINICAL TRIAL: NCT05624645
Title: Efficacy of a Non-invasive Pelvic Floor Muscle Trainer for Treatment of Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX-001
Record Dates: First submitted 2022-10-30; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence; Pelvic Floor Disorders
Keywords: stress urinary incontinence; pelvic floor disorders
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pelex Upp (Experimental): In this arm, all patients received the device for use in treatment of stress urinary incontinence.
  Interventions: Device: Pelex Upp

INTERVENTIONS:
Device: Pelex Upp — Patients were given the Pelex Upp is a non-invasive device that is designed to guide a user through personalized pelvic floor strengthening exercises. Patients used device for four weeks to treat stress urinary incontinence

SUMMARY:
The goal of this clinical trial is to assess the efficacy and usability of the electromyography component of the company's pelvic health product in a patient population with stress urinary incontinence. The main questions it aims to answer are:

Does treatment with the device under study improve symptoms of stress urinary incontinence as measured by the ICIQ?

Participants will be given one of the devices under study, in addition to educational materials on use of the device, and a treatment schedule. Participants will perform a standardized biofeedback-mediated pelvic floor muscle training program with the study device 10 minutes a day, five times a week for 4 weeks. There will be a mid-study check in to assure all devices are functioning appropriately. At the end of the study, participants will complete a post-treatment urinary incontinence symptom questionnaire(ICIQ).

DETAILED DESCRIPTION:
This will be a prospective cohort study of women > 18 years of age with symptoms of stress urinary incontinence, recruited via an online recruitment tool.

After screening, patients meeting inclusion criteria will be given a study brochure, and then given instructions on how to indicate desire to participate in the study. The patient will then be contacted for study participation, including explanation of study and details and completion of Informed Consent. Participants will then complete a pre-treatment urinary incontinence symptom questionnaire(ICIQ).

After completion of the above, the participants will then be given one of the devices under study, in addition to educational materials on use of the device, and a treatment schedule. Participants will perform a standardized biofeedback-mediated pelvic floor muscle training program with the study device 10 minutes a day, five times a week for 4 weeks. There will be a mid-study check in to assure all devices are functioning appropriately. At the end of the study, participants will complete a post-treatment urinary incontinence symptom questionnaire(ICIQ).

Endpoint of the study will be change in stress urinary incontinence symptoms as measured by the ICIQ. The ICIQ will be collected at 2 time points: before study entry, and at study close.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Documented symptoms of predominantly stress urinary incontinence as determined by the ICIQ questionnaire

Exclusion Criteria:

* History of pelvic or lower back surgery

Pregnancy or less than 12 months post partum

History of physician-supervised PFMT

History of Kegel exercises greater than once a month

History of prior operative delivery

Self-reported history of pelvic organ prolapse stage II or greater

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Change in stress urinary incontinence symptoms | 4 weeks
  Patients were given the ICIQ-UI SF, the standard assessment tool for stress and urge urinary incontinence, both before initiation and at the end of study. The difference between the two scores was then assessed to determine whether an change in stress urinary incontinence symptoms occurred after use of the device.
  ICIQ is the International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form is a four question survey to "evaluate the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women." It has a maximum and minimum score of 21 and 0 respectively. Higher scores reflect more significant urinary incontinence symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Wiygul, M.D., Principal Investigator — Pelex
Locations (1):
- Pelex, Little Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgio KL, Locher JL, Goode PS, Hardin JM, McDowell BJ, Dombrowski M, Candib D. Behavioral vs drug treatment for urge urinary incontinence in older women: a randomized controlled trial. JAMA. 1998 Dec 16;280(23):1995-2000. doi: 10.1001/jama.280.23.1995. PMID 9863850
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Chong EC, Khan AA, Anger JT. The financial burden of stress urinary incontinence among women in the United States. Curr Urol Rep. 2011 Oct;12(5):358-62. doi: 10.1007/s11934-011-0209-x. PMID 21847532
- [Background] Seyyedi F, Rafiean-Kopaei M, Miraj S. Comparison of the Effects of Vaginal Royal Jelly and Vaginal Estrogen on Quality of Life, Sexual and Urinary Function in Postmenopausal Women. J Clin Diagn Res. 2016 May;10(5):QC01-5. doi: 10.7860/JCDR/2016/17844.7715. Epub 2016 May 1. PMID 27437306
- [Background] Berghmans LC, Hendriks HJ, Bo K, Hay-Smith EJ, de Bie RA, van Waalwijk van Doorn ES. Conservative treatment of stress urinary incontinence in women: a systematic review of randomized clinical trials. Br J Urol. 1998 Aug;82(2):181-91. doi: 10.1046/j.1464-410x.1998.00730.x. PMID 9722751
- [Background] KEGEL AH. Progressive resistance exercise in the functional restoration of the perineal muscles. Am J Obstet Gynecol. 1948 Aug;56(2):238-48. doi: 10.1016/0002-9378(48)90266-x. No abstract available. PMID 18877152
- [Background] Pages IH, Jahr S, Schaufele MK, Conradi E. Comparative analysis of biofeedback and physical therapy for treatment of urinary stress incontinence in women. Am J Phys Med Rehabil. 2001 Jul;80(7):494-502. doi: 10.1097/00002060-200107000-00006. PMID 11421517
- [Background] Burns PA, Pranikoff K, Nochajski TH, Hadley EC, Levy KJ, Ory MG. A comparison of effectiveness of biofeedback and pelvic muscle exercise treatment of stress incontinence in older community-dwelling women. J Gerontol. 1993 Jul;48(4):M167-74. doi: 10.1093/geronj/48.4.m167. PMID 8315230
- [Background] Dumoulin C, Bourbonnais D, Morin M, Gravel D, Lemieux MC. Predictors of success for physiotherapy treatment in women with persistent postpartum stress urinary incontinence. Arch Phys Med Rehabil. 2010 Jul;91(7):1059-63. doi: 10.1016/j.apmr.2010.03.006. PMID 20537314
- [Background] Herderschee R, Hay-Smith EJ, Herbison GP, Roovers JP, Heineman MJ. Feedback or biofeedback to augment pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD009252. doi: 10.1002/14651858.CD009252. PMID 21735442
- [Background] Glazer HI, Laine CD. Pelvic floor muscle biofeedback in the treatment of urinary incontinence: a literature review. Appl Psychophysiol Biofeedback. 2006 Sep;31(3):187-201. doi: 10.1007/s10484-006-9010-x. PMID 16983505
- [Background] Moroni RM, Magnani PS, Haddad JM, Castro Rde A, Brito LG. Conservative Treatment of Stress Urinary Incontinence: A Systematic Review with Meta-analysis of Randomized Controlled Trials. Rev Bras Ginecol Obstet. 2016 Feb;38(2):97-111. doi: 10.1055/s-0035-1571252. Epub 2016 Jan 29. PMID 26883864
- [Background] Barnes KL, Cichowski S, Komesu YM, Jeppson PC, McGuire B, Ninivaggio CS, Dunivan GC. Home Biofeedback Versus Physical Therapy for Stress Urinary Incontinence: A Randomized Trial. Female Pelvic Med Reconstr Surg. 2021 Oct 1;27(10):587-594. doi: 10.1097/SPV.0000000000000993. PMID 33208658
- [Background] Rosenblatt P, McKinney J, Rosenberg RA, Iglesias RJ, Sutherland RC, Pulliam SJ. Evaluation of an accelerometer-based digital health system for the treatment of female urinary incontinence: A pilot study. Neurourol Urodyn. 2019 Sep;38(7):1944-1952. doi: 10.1002/nau.24097. Epub 2019 Jul 16. PMID 31310369
- [Background] Washington BB, Raker CA, Sung VW. Barriers to pelvic floor physical therapy utilization for treatment of female urinary incontinence. Am J Obstet Gynecol. 2011 Aug;205(2):152.e1-9. doi: 10.1016/j.ajog.2011.03.029. Epub 2011 Mar 22. PMID 21620356

DOCUMENTS (2):
  • Study Protocol (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT05624645/Prot_000.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT05624645/ICF_001.pdf